CLINICAL TRIAL: NCT06459154
Title: The Effectiveness of Mixed Reality as Interventional Tool for the Improvement on Quality of Life for People With Parkinson´s Disease. Randomized Control Trial
Brief Title: The Effectiveness of Mixed Reality as Interventional Tool for the Improvement on Quality of Life for People With Parkinson´s Disease.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nicosia (Other)
Responsible Party: Principal Investigator, Elena Papamichael, PhD Candidate in Physiotherapy, University of Nicosia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ΕΕΒΚ/ΕΠ/2023/07
Record Dates: First submitted 2024-05-15; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
Keywords: PD; Mixed Reality; Physiotherapy; QOL; Motivation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Parallel assignment of Randomized Control Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mixed Reality interventional Group (Experimental)
  Interventions: Other: Mixed Reality; Other: Traditional Physiotherapy
- Traditional Physiotherapy Group (Experimental)
  Interventions: Other: Mixed Reality; Other: Traditional Physiotherapy
- Placebo group (Placebo Comparator)
  Interventions: Other: Mixed Reality; Other: Traditional Physiotherapy

INTERVENTIONS:
Other: Mixed Reality — The experimental group MR will use the mixed reality project involving activities in a supermarket. MR HoloLens2 glasses will be used to conduct the program. The technological equipment that will be used will allow the provision of visual and auditory stimuli. The program presents 5-10 different objects found in a supermarket, where you need, as you walk, to collect them within a mixed environment. This program offers coordination activities, posture, cognitive activities and balance exercises. The mixed reality program lasts 30 minutes, with a frequency of 3 times a week for 12 weeks.
Other: Traditional Physiotherapy — The group of traditional physiotherapy follows the guidelines of EPDA. Specifically, the program will be 35-40 minutes long, 3 times a week for 12 weeks. The program includes 5 minutes warm up, 10 minutes resistance exercises, 10 minutes of balance exercises and stretching.

SUMMARY:
Parkinson's disease is a chronic, neurodegenerative disease of unknown cause, affecting elderly people over the age of 60. It is the second most common neurodegenerative disease, presenting psychomotor signs and symptoms that lead to impaired functionality and quality of life in affected individuals. Mixed reality involves the delivery of digital stimuli in real time and space through spatial mapping using glasses, safely providing multiple iterations to carry out daily activities.

Through this tool and in collaboration with technologically skilled mixed reality developers, the software for the rehabilitation program to be applied to Parkinson's disease patients was also developed.

The main objective of this clinical study is to examine the effect of a mixed reality program compared to a traditional physiotherapy program on quality of life and motivation for the participation of people with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a chronic, neurodegenerative disease of unknown cause, affecting elderly people over the age of 60. It is the second most common neurodegenerative disease, presenting psychomotor signs and symptoms that lead to impaired functioning and quality of life in affected individuals. Mixed reality involves the delivery of digital stimuli in real time and space through spatial mapping using glasses, safely providing multiple iterations to carry out daily activities.

Through this tool and in collaboration with technologically skilled mixed reality developers, the software for the rehabilitation program to be applied to Parkinson's disease patients was also developed.

The main objective of this clinical study is to examine the effect of a mixed reality program compared to a traditional physiotherapy program on quality of life and motivation for the participation for people with Parkinson's disease.

The study will be divided into two phases, the first of which includes the translation and adaptation of the Intrinsic Motivation Inventory (IMI) questionnaire, which assesses motivation and is not available in Greek, and will be used in 300 healthy subjects to assess its psychometric characteristics.

The second phase of the clinical trial is a parallel, blinded, randomized study involving 45 patients.

This study will provide the opportunity to use innovative equipment that offers multiple stimuli increasing the interactivity of the participants to perform functional activities. This research is the first clinical study in Cyprus that will apply the reported rehabilitation tool aiming to improve and evaluate the quality of life, functionality and motivation of people with Parkinson's disease. Moreover, it enables the development of cognitive and motor rehabilitation by increasing the interaction of the individual with the environment and facilitating the completion of treatment goals.

The research using mixed reality and through a comparative process with traditional physiotherapy, aims to provide valid and reliable data to the general public and health scientists, facilitating the selection of appropriate means to provide a holistic treatment plan.

Translated with DeepL.com (free version)

ELIGIBILITY:
For the first interventional phase:

Inclusion Criteria:

1. Male and female over 18 years old 2. Persons with independent gait 3. Normal cognitive ability 5. Greek Native language

Exclusion Criteria:

1. Presence of neurological disease
2. Presence of uncontrolled diseases of the circulatory system
3. History of musculoskeletal surgery in the last 6 months
4. Use of a walking aid
5. Partial or total blindness

For the second interventional phase:

Inclusion Criteria:

1. Male and female over 60 years old
2. Persons with independent gait
3. Normal cognitive ability

5. Greek Native language

Exclusion Criteria:

1. Presence of neurological disease
2. Presence of uncontrolled diseases of the circulatory system
3. History of musculoskeletal surgery in the last 6 months
4. Use of a walking aid
5. Partial or total blindness

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2025-02-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
EuroQol 5 Dimension 5 Level | baseline, 4weeks follow up
  Measurement of quality of life. Likert scoring style (1-5) where higher scores represent worse state of quality of life
The Short Form (12) Health Survey | baseline, 4weeks follow up
  Measurement of quality of life: The scores ranged from 0 to 100, where higher scores representing better quality of life

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory | baseline, 4weeks follow up
  Measurement of intrinsic motivation: That contains 7 subcategories with average score from 1 to 7. Higher scores indicating better motivation
Mini Balance Evaluation Systems Test | baseline, 4weeks follow up
  Measurement of functionality and Balance: The scale's scores ranging from 0 to 28, where higher scores represent better functionality
Multidirectional Reach Test | baseline, 4weeks follow up
  Measurement of balance and functionality: Is the only scale that includes cm for the measurement of distance. Most healthy people present 25cm. People who present less than 18cm, indicates limitations on functional balance
Nine-Hole Peg Test | baseline, 4weeks follow up
  Measurement of fine motor skills and functionality: The test scores are based on the average duration of four trials. Healthy females present 17.9-19.6 second and males 19-20.6 seconds. Higher average duration indicates limited fine mobility

CONTACTS AND LOCATIONS:
Overall Officials: Elena Papamichael, PhD Cand, Principal Investigator — University of Nicosia
Locations (1):
- University of Nicosia, Nicosia, Engomi, Cyprus